CLINICAL TRIAL: NCT03129217
Title: The Validity of Maximal Diaphragm Thickening Fraction to Measure Diaphragm Function in Mechanically Ventilated Patients
Acronym: SNIFF III
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ewan Goligher, Clinical Associate, University Health Network, Toronto
Other Study IDs: 15-9644-AE
Record Dates: First submitted 2017-04-05; First posted 2017-04-26 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Diaphragm Injury; Weaning Failure; Mechanical Ventilation Complication
Keywords: Diaphragm function; Acute respiratory failure; Weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients weaning from mechanical ventilation

SUMMARY:
This study is designed to determine whether maximal diaphragm thickening fraction measured by ultrasound during volitional maximal inspiratory efforts is a valid measure of diaphragm function in mechanically ventilated patients.

DETAILED DESCRIPTION:
Classically, assessing diaphragm function requires direct measurements of transdaphragmatic pressure generation. A critical requirement for valid measurements is a maximal volitional patient effort. An alternative is to standardize the stimulus to the diaphragm using magnetic twitch stimulation fo the phrenic nerve. This is the gold standard technique for diaphragm function measurement in the respiratory physiology laboratory.

Twitch measurements require technical expertise and expensive equipment; this technique is therefore basically limited to the laboratory. Bedside ultrasonography has been proposed as a method for measuring diaphragm function by assessing the thickening of the muscle during a maximal inspiratory effort. In order to achieve a maximal volitional effort in mechanically ventilated patients, several methods may be employed: coached maximal efforts, coached sniffing, and transient airway occlusion to stimulate respiratory drive (Marini maneuver).

The investigators are evaluating the validity of diaphragm functional assessment using bedside ultrasound in combination with coached efforts/sniffing/Marini maneuver against the gold standard technique: twitch transdiaphragmatic pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) with acute respiratory failure receiving invasive mechanical ventilation via endotracheal tube or tracheostomy
* Patients who meet readiness-to-wean criteria (triggering the ventilator; FiO2 ≤ 50%; PEEP ≤ 8 cm H20; hemodynamic stability)

Exclusion Criteria:

* Contraindication to phrenic nerve stimulation (chest tube; cardiac pacemaker or implanted defibrillator; cervical implants; use of neuromuscular blocking agents within the 24 hours preceding the first diaphragm assessment (with the exception of succinylcholine used during rapid-sequence induction of anaesthesia for intubation); cervical spine injury; known pregnancy)
* Patients experiencing an acute exacerbation of an obstructive lung disease (chronic obstructive pulmonary disease (COPD), asthma, bronchiectasis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with acute respiratory failure requiring invasive mechanical ventilation who meet readiness-to-wean criteria.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Maximal diaphragm thickening fraction | On day of study
  Diaphragm ultrasound to measure thickening fraction

CONTACTS AND LOCATIONS:
Overall Officials: Ewan C Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to make data available to other researchers.